CLINICAL TRIAL: NCT05639205
Title: Shaping Care Home COVID-19 Testing Policy: A Pragmatic Cluster Randomised Controlled Trial of Asymptomatic Testing Compared to Standard Care in Care Home Staff.
Brief Title: Shaping Care Home COVID-19 Testing Policy
Acronym: VIVALDI-CT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CTU/2022/405
Record Dates: First submitted 2022-12-02; First posted 2022-12-06 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
Keywords: Lateral Flow Device
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): LFD testing for Covid-19 with sickness support payment. Care providers will receive funding to reimburse the costs of employing agency staff to cover sickness absence in asymptomatic staff who test positive for COVID.
  Interventions: Diagnostic Test: Lateral Flow Device
- Arm B (No Intervention): Usual Care

INTERVENTIONS:
Diagnostic Test: Lateral Flow Device — Regular asymptomatic staff testing with a Lateral Flow Device including support payments if unwell.
  Arms: Arm A

SUMMARY:
The goal of this interventional study is to investigate whether continued use of regular asymptomatic testing in staff is a feasible, effective and cost-effective strategy to reduce the impact of COVID-19 in care homes.

The trial aims to quantify the benefits and harms of regular asymptomatic testing in care home staff to inform policy. The rationale for regular asymptomatic testing is that it may reduce the risk of severe disease in residents and the frequency/severity of outbreaks.

Participants (care home staff) will perform regular asymptomatic tests for Covid-19. Should they test positive they will be required to refrain from working and be provided with sick pay.

Care providers will be reimbursed for the costs of employing agency staff to cover staff sickness absence that results directly from the trial.

DETAILED DESCRIPTION:
To date the evidence based underpinning elements of the intervention has been developed through engagement work with the National Care Forum, senior managers of care homes and three stakeholder events with front-line care home staff. It will be finalised through a series of further workshops. These workshops will 1) consolidate existing insights into routine testing gleaned through past experiences in the COVID-19 pandemic; 2) discuss the intervention prototype; 3) operationalise it in ways which are likely to be acceptable and appropriate within the sector.

The testing intervention will comprise of four modules that will be delivered in combination. Module 1: support payments for staff to enable them to self-isolate when unwell. Module 2: Branding and messaging around testing to promote engagement with testing. Module 3: Accessing training, protocols and planning. Module 4: Regular asymptomatic staff testing for COVID-19 using LFDs.

Asymptomatic testing will be in addition to symptomatic testing for staff and residents, which is standard policy for all care homes in England.

Providers will also receive funding to reimburse costs associated with employing agency staff to cover sickness absence for asymptomatic staff who test positive in the trial.

Non-intervention care home residents and staff will be subject to the testing policy that is in place nationally at the time of the trial. Care home staff in control homes will not receive support payments (Module 1) and testing in control homes will not be supported by branding or messaging (Module 2). The degree to which training and testing protocols are already in place in control homes (Module 3) will be investigated in the stakeholder workshops.

ELIGIBILITY:
Inclusion Criteria:

* Only care home staff are eligible to participate in the testing intervention. This includes temporary (agency) staff with no restrictions i.e. catering staff, administrative staff, maintenance staff, in addition to those in a resident-facing role.
* All care home staff, residents, visitors and relatives are eligible to participate in interviews undertaken as part of the process evaluation.
* All care home residents at participating home are eligible for data collection and analysis of the outcomes specified.

Exclusion Criteria:

* Visitors, residents and relatives are not eligible to take part in the testing intervention.
* Staff who visit the care home to provide care but are not employed by the care home e.g. GPs, health visitors are not eligible to take part in either the interviews or the testing intervention.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 4 months
  The primary outcome is the incidence of COVID-19 related hospital admissions in residents, defined as admissions with a relevant ICD-10 codes (COVID hospitalisations to be defined as any hospital admission record with a primary or secondary ICD10 code of 'U071') and/or admissions in residents who test positive for COVID-19 within 24h following admission or in the 7 days before hospital admission. This has been selected because it is the most important outcome for policymakers.

SECONDARY OUTCOMES:
Incidence rate of hospital admissions | 4 months
  Incidence rate of hospital admissions (all-cause) in residents for non-elective care, measured as events per 100,000 person-days of follow-up over the duration of the trial
Incidence rate of COVID-associated mortality in residents | 4 months
  Incidence rate of COVID-associated mortality in residents, measured as events per 100,000 person-days of follow-up over the duration of the trial.
  COVID-associated mortality will be defined as death within 28 days of a positive SARS-CoV-2 test and/or COVID-19 recorded as primary or secondary cause of death on the death certificate (using ICD-10 coding).
Incidence of all-cause mortality in residents | 4 months
  Incidence of all-cause mortality in residents, measured as events per 100,000 person-days of follow-up over the duration of the trial
Testing uptake in staff | Once per week for 4 months
  Testing uptake in staff, measured as proportion of staff at each home participating in testing during each week of the trial
Prevalence of SARS-CoV-2 among staff who test | Once per week for 4 months
  Prevalence of SARS-CoV-2 among staff who test, measured as proportion of staff with positive test result among those with at least one test recorded during each week of the trial
Incidence rate of SARS-CoV-2 infections detected in residents | 4 months
  Incidence rate of SARS-CoV-2 infections detected in residents, measured as events per 100,000 person-days of follow-up over the duration of the trial
Incidence rate of home-level outbreaks | 4 months
  Incidence rate of home-level outbreaks, measured as events per 1000 days of follow-up over the duration of the trial
Duration of outbreaks | 4 months
  Duration of outbreaks, measured as days from first to last case within outbreaks occurring within the trial period
Incidence rate of care home closures due to outbreaks | 4 months
  Incidence rate of care home closures due to outbreaks, measured as events per 1000 days of follow-up over the duration of the trial
Staff sick | Once per week for 4 months
  Proportion of staff per home who are off sick at each home during each week of the trial
Agency staff filled shifts | Once per week for 4 months
  Proportion of all shifts filled by agency staff at each home during each week of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Laura Shallcross, Professor, Principal Investigator — UCL

IPD SHARING:
Plan to Share IPD: Undecided
The data-sharing plans for the current study are still to be confirmed and will be made available at a later date.

REFERENCES:
- [Derived] Stirrup O, Blackstone J, Cullen-Stephenson I, Fenner R, Adams N, Leiser R, Krutikov M, Azmi B, Freemantle N, Gordon A, Regan M, Knapp M, Gosce L, Henderson C, Hopkins S, Verma A, Cassell J, Cadar D, Fowler T, Copas A, Flowers P, Shallcross L. VIVALDI-CT shaping care home COVID-19 testing policy: A pragmatic cluster randomised controlled trial of asymptomatic testing compared to standard care in care home staff. PLoS One. 2025 Jul 2;20(7):e0324908. doi: 10.1371/journal.pone.0324908. eCollection 2025. PMID 40601586